CLINICAL TRIAL: NCT07257861
Title: Interest of Continuous Subcutaneous Apomorphine in Parkinsonian Patients at the End of Life
Acronym: OPTIDOM
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Collaborators: Fédération Francaise d'Hospitalisation à Domicile (FNEHAD) (Unknown); France Développement Electronique (FDE) (Unknown)
Responsible Party: Sponsor
Other Study IDs: CHUO-2025-02
Record Dates: First submitted 2025-09-18; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Parkinson Disease
Keywords: Apomorphine; Parkinson; End of life
MeSH Terms: conditions — Parkinson Disease; Death | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Parkinson patients: Parkinsonian patients in HH will receive an apomorphine pump as part of their routine care.
  Questionnaires will be completed at D0, D2, D4, D6, D12, D18, D24, D30 and D45. The questionnaires used will be
  * UPDSR III: rigidity
  * Algoplus
  * Richmond Scale (RASS)
  * Likert scale Entourage before/after
  * Likert scale Caregivers before/after
  * Zarit scale
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Parkinsonian patients in HH will receive an apomorphine pump as part of their routine care.
  Questionnaires will be completed at D0, D2, D4, D6, D12, D18, D24, D30 and D45. The questionnaires used will be
  * UPDSR III: stiffness
  * Algoplus
  * Richmond Scale (RASS)
  * Likert scale Entourage before/after
  * Likert scale Caregivers before/after
  * Zarit scale

SUMMARY:
Care for Parkinson's patients at the end of life is far from optimal, particularly due to specificities linked to the disease itself, often unknown to non-specialists.

A study carried out at the CHU Rennes on data covering the period 2006-2018 showed that only 132 patients died in this hospital, two-thirds of whom came from home. In 42% of cases, antiparkinsonian treatment was stopped before death without specialist advice (palliative or neurological), with the corollary of the appearance of a dopaminergic withdrawal syndrome (or pseudo-neuroleptic malignant syndrome) in a high proportion of these patients. Neuroleptic pseudo-malignant syndrome is a major cause of discomfort. If left untreated, it can precipitate death in particularly distressing conditions for the patient, his or her family and caregivers.

The Rennes study also suggests that Parkinson's patients rarely die in hospital. In fact, work carried out by FNEHAD on data for 2022 showed that 1,800 Parkinson's patients were cared for in HAH in France during that same year, mainly for palliative care or heavy nursing reasons. Half of these patients died.

End-of-life management of Parkinson's disease therefore requires local clinical and pharmacological expertise. A recent observational study suggests that the use of a subcutaneous apomorphine pump brings substantial benefits in terms of clinical comfort, both motor and non-motor, as well as relief for family and friends, easier nursing care for the nursing team, and in some cases, renewed communication.

Such care can be provided in the home, and must necessarily be multidisciplinary, combining palliative expertise, provided by Home Hospitalization (HH) teams, with technical and Parkinson's expertise, provided by Home Healthcare Providers (HHPs) experienced in managing the apomorphine pump, in liaison with the referral team.

ELIGIBILITY:
Inclusion Criteria:

1. Person (or trusted person/relative if patient is unable) who has agreed to participate in the study
2. Patient of legal age
3. Advanced Parkinson's disease with apomorphine pump indication
4. Use of HH for palliative reasons
5. Loss of orality (discontinuation of oral treatments)
6. Hoehn &Yahr score in OFF = 5 (bilateral and axial symptoms in the absence of levodopa)

Exclusion Criteria:

1. Apomorphine pump already in use
2. Opposition to the introduction of an apomorphine pump
3. Protected person (under guardianship or curatorship)
4. Person under court protection
5. Persons deprived of liberty
6. Persons not affiliated to a social security scheme
7. Pregnant or breast-feeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parkinsonian patients treated in HH.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Rigidity | Day 0
  measured by the specific sub-section of rigidity of the internationally recognized UPDRS 3 scale validated in French. This criterion will be assessed before the apomorphine pump is installed and 6 days afterwards.
  The 5 items are scored from 0 to 4, so the total score ranges from 0 to 20.
Rigidity | Day 6
  measured by the specific sub-section of rigidity of the internationally recognized UPDRS 3 scale validated in French. This criterion will be assessed before the apomorphine pump is installed and 6 days afterwards.
  The 5 items are scored from 0 to 4, so the total score ranges from 0 to 20.

SECONDARY OUTCOMES:
Change in analgesic consumption | Day 45
  Change in analgesic consumption will be recorded at Day 0, 2, 4, 6, 12, 18, 24, 30 and Day 45 and will be evaluated at the end of the study
Change in alertness and agitation levels | Day 45
  It will be will be evaluated by the Richmond Scale, from + 4 to -4 with +4 for very combative patient and -4 for unresponsive patient.
Change in communication with the care team and relatives | Day 45
  It will be evaluated with the Lickert scale for care team that assesses the patient's communication ability from -3 to +3 with -3 for greatly aggravated and +3 for greatly improved
Change in nursing care | Day 45
  It will be evaluated with the Lickert scale for caregivers that assesses the level of quality of nursing care. from -3 to +3 with -3 for greatly aggravated and +3 for greatly improved
Change in caregiver burden | Day 0, 2, 6, 18, 30 and Day 45
  It will be evaluated with Zarit scale . The total score is the sum of the scores obtained for each of the 22 items, ranging from 0 to 88. A score of 20 or less indicates a low or no burden; a score between 21 and 40 indicates a mild burden; a score between 41 and 60 indicates a moderate burden; a score above 60 indicates a severe burden.
Proportion of nausea/vomiting | Day 0, 2, 4, 6, 12, 18, 24, 30 and Day 45
Proportion of hypotension | Day 0, 2, 4, 6, 12, 18, 24, 30 and Day 45
Proportion of skin condition related to apomorphine | Day 0, 2, 4, 6, 12, 18, 24, 30 and Day 45
Proportion of hallucinations | Day 0, 2, 4, 6, 12, 18, 24, 30 and Day 45